CLINICAL TRIAL: NCT06937983
Title: Optimised Decrement Evoked Potential (DeEP) Mapping to Guide Ventricular Tachycardia (VT) Ablation in Patients With Structural Heart Disease VT
Acronym: Opto-DeEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD636723
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Structural Heart Disease
Keywords: Ventricular Tachycardia; Decrementing Evoked Potential mapping; Optimisation parameters; Clinical Applicability
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimised DeEP-guided ablation (Experimental): DeEP mapping in VT ablation.
  Interventions: Procedure: Optimised DeEP-guided ablation

INTERVENTIONS:
Procedure: Optimised DeEP-guided ablation — Optimised decrement evoked potential (DeEP) mapping in VT ablation.

SUMMARY:
Ventricular tachycardia (VT) is a life-threatening heart rhythm disorder. Special pacemakers called implantable cardiac defibrillators (ICDs) help treat VT episodes, however they do not prevent the VT episodes from occurring. Catheter ablation for VT is a minimally-invasive and established procedure for preventing VT recurrence. This involves placing wires in the heart to find the diseased areas that are responsible for the VT episodes. The diseased areas are shown on computer-generated maps and are later removed via controlled tissue heating (ablation). A major challenge during the VT ablation procedure is locating the diseased area responsible for the VT episodes. Several methods have been described to locate the diseased heart area, however these methods are not always effective.

In this study, we aim to improve the identification of the diseased heart areas responsible for the VT episodes using a novel method. Our research group have developed, tested and peer-reviewed this improved method of locating diseased areas by looking for signals called decrementing evoked potentials (DeEPs). Ablation will target DeEPs shown on the computer-generated maps. We will assess if VT can be triggered at the end of the procedure. Patients will be monitored over 12 months to see if ablation of DeEPs leads to a reduction in VT episodes. We aim to recruit 77 patients with established heart disease of any cause, who have suffered VT episodes with ICDs. Suitable patients will be identified and recruited from inpatient and outpatient settings. A quality-of-life questionnaire will be completed by patients before and after the ablation procedure. The procedure will be performed as routine standard of care, in the cardiac catheter laboratory across multiple recruiting cardiac centres in the UK providing well established VT ablation service.

Overall, this study will contribute towards developing refined VT ablation techniques, aiming to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients with cardiac implantable electronic devices (CIED) (e.g. pacemakers, cardiac resynchronisation therapy (CRT) devices, implantable cardioverter defibrillator (ICD) devices)
* Eligible for VT ablation as part of standard care (urgent or elective)
* Ischaemic heart disease and prior myocardial infarction (MI) (using the international definition of MI: Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non-ischemic cause with documentation of prior ischaemic injury) OR other structural heart disease (such as: arrhythmogenic cardiomyopathy (ACM), or dilated cardiomyopathy (DCM), or hypertrophic cardiomyopathy (HCM), or sarcoidosis, or myocarditis).
* VT ablation to be performed using Abbott intracardiac mapping catheter and Ensite intracardiac mapping system, using radiofrequency (RF) energy source.

Exclusion Criteria:

* Lacks capacity to provide informed consent
* New York Heart Association (NYHA) class IV heart failure
* Life expectancy of less than 12 months
* Implanted with a ventricular assist device
* Presence of mobile intracardiac thrombus
* Reversible cause of VT
* Women who are pregnant or nursing
* Both mechanical aortic and mitral valves
* Enrolment in a concurrent interventional clinical study that in the judgement of the investigator would increase risk to the patient or deem the patient inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-12-03 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
To determine acute success rate post Opto-DeEP mapping-guided VT ablation. | From the start to the end of the VT ablation procedure.
  Number of patients with non-inducible VT acutely after optimised DeEP map-guided ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised data will be shared on request to the Sponsor and Chief Investigator.